CLINICAL TRIAL: NCT06663605
Title: A Phase 1, Double-Blind, Placebo-Controlled, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of PALI-2108 in Healthy Volunteers and Open-Label Study of a Patient Cohort With Ulcerative Colitis
Brief Title: Phase 1 Study Evaluating PALI-2108 in Healthy Volunteers and Ulcerative Colitis Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Palisade Bio (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBI-2108-101
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis (UC); Healthy Volunteer
Keywords: Phase 1 for PALI-2108 in Healthy Volunteers and UC patients; Ulcerative colitis; PALI-2108
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Phase 1 a/b Double-Blind, Placebo-Controlled, Randomized Single Ascending Dose (SAD)/Multiple Ascending Dose (MAD), Food Effects (FE) crossover and Open-Label Ulcerative Colitis patient cohort study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PALI-2108 (Experimental): Part A - Single Ascending oral doses of PALI-2108 in healthy adult subjects. Part B - Single oral dose crossover of PALI-2108 in healthy adult subjects. Part C - Multiple Ascending oral Doses of PALI-2108 in healthy adult subjects. Part D - (open-label) Multiple oral Doses of PALI-2108 in Ulcerative Colitis patients.
  Interventions: Drug: PALI-2108
- PALI-2108 Placebo (Placebo Comparator): Part A - Single Ascending oral Dose of matching placebo in healthy adult subjects. Part B - Single Ascending oral Dose of matching placebo crossover of PALI-2108 in healthy adult subjects. Part C - Multiple Ascending oral Doses of matching placebo in healthy adult subjects. Part D - (open-label) Multiple Ascending oral Doses of matching placebo in Ulcerative Colitis patients.
  Interventions: Drug: PALI-2108 Placebo

INTERVENTIONS:
Drug: PALI-2108 — Oral dose
  Other Names: PALI-2108 active drug
  Arms: PALI-2108
Drug: PALI-2108 Placebo — Oral dose
  Arms: PALI-2108 Placebo

SUMMARY:
PALI-2108 is a new oral medication designed to treat ulcerative colitis (UC) by targeting the intestines. It works as a phosphodiesterase-4 (PDE4) inhibitor prodrug, meaning it becomes active only after being processed by bacteria in the colon. This targeted approach reduces the risk of side effects that can occur with other medications that affect the entire body.

Recent studies have shown that patients with active UC, especially those with moderate to severe symptoms, have higher levels of PDE4 and related biomarkers. These biomarkers are linked to the severity of their disease, suggesting that inhibiting PDE4 could help manage UC effectively.

The goal of this Phase 1 study is to evaluate the safety, tolerability, and how the body processes (pharmacokinetics) and responds to (pharmacodynamics) PALI-2108 in healthy volunteers. Although there are already PDE4 inhibitors on the market, PALI-2108 is a completely new compound that has not been tested in humans before. The study will involve two parts: first, participants will receive single doses of the drug, and then, in the second part, they will take it twice a day for seven days.

The twice-daily dosing schedule is designed to maximize drug exposure in the colon. The investigators will also investigate how food affects the drug's absorption.

Additionally, a small group of stable UC patients will be included in the study. These patients will also take PALI-2108 for seven days, allowing us to compare the safety and drug processing between healthy individuals and those with UC. The investigators will monitor important health markers and conduct tests on colon tissue to see how well the drug works and if it causes any changes in the tissue.

Including UC patients early in this research is important for understanding how the drug performs in real-world conditions. This data will help refine our approach to identify which patients might benefit most from PALI-2108 in future studies.

Overall, this study aims to gather crucial information about PALI-2108's safety and effectiveness, paving the way for new treatment options for patients with ulcerative colitis.

DETAILED DESCRIPTION:
PALI-2108 is a novel synthetic prodrug designed to function as an intestinally activated phosphodiesterase-4 (PDE4) inhibitor, with a unique galactose sugar moiety linked by a beta 1,4 bond that enhances its targeted delivery within the colon. This innovative formulation minimizes systemic exposure and potential central nervous system (CNS) mediated toxicity by being cleaved by colonic bacterial enzyme β-glucuronidase, thus releasing the active PDE4 inhibitor directly in the colonic tissue. This mechanism is particularly advantageous in treating conditions like ulcerative colitis (UC), where localized treatment can enhance safety and efficacy.

Recent proprietary bioinformatics analyses indicate that patients with active UC, especially those with moderate to severe disease, exhibit significantly elevated levels of PDE-4 and PDE-4 related transcriptional biomarkers. These biomarkers have been found to correlate with established markers of UC disease activity and severity, such as the Mayo score. This highlights the potential role of PDE-4 inhibition in managing UC, making PALI-2108 a promising candidate for further investigation.

The primary aim of this single-center Phase 1 study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of PALI-2108 in healthy volunteers. Although several PDE-4 inhibitors have received market approval, but not in Ulcerative Colitis, PALI-2108 represents a new chemical entity that has not been previously administered to humans. The study will consist of single ascending dose (SAD) cohorts followed by multiple ascending dose (MAD) cohorts, with participants receiving twice-daily (BID) dosing for seven consecutive days. This BID regimen is designed to optimize colonic exposure to the active PDE4 inhibitor.

In addition to healthy volunteers, a small cohort of stable moderate to severe UC patients will be included in the study. These patients, who will be under standard care, will also receive BID dosing for seven days. Comprehensive safety monitoring and similar PK evaluations will be conducted in this cohort. Biomarkers, including high sensitivity C-reactive protein (hsCRP) and fecal calprotectin (CalPro), along with colonic tissue histological assessments, will be employed to provide further insights into the drug's effects. The analysis of colon tissue will include the study drug and metabolite levels, PDE4 expression, and related PD biomarkers, which are crucial for understanding the drug's mechanism and efficacy.

This early inclusion of UC patients is strategic, allowing for the correlation of PK/PD profiles between healthy volunteers and UC subjects. It also enables close monitoring of safety within a controlled clinical pharmacology unit. The comprehensive data gathered will support Palisade Bio's Precision Medicine Strategy, aimed at identifying patient responders for future clinical studies. Overall, the study of PALI-2108 has the potential to advance therapeutic options for UC, emphasizing localized treatment and improved patient safety.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects and patients:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. If male, meets one of the following criteria:

   1. Is able to procreate and agrees to use one of the accepted contraceptive regimens and not to donate sperm from the first study drug administration to at least 90 days after the last study drug administration. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository) Or
   2. Is unable to procreate; defined as surgically sterile (eg, has undergone a vasectomy at least 180 days prior to the first study drug administration)
4. If female, is of non-childbearing potential and meets one of the following criteria:

   1. Is surgically sterile (ie, has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) Or
   2. Is in a postmenopausal state:

      * At least 1 year without menses and without an alternative medical condition prior to the Screening visit and follicle stimulating hormone [FSH] levels ≥ 40 mIU/mL at Screening Or
      * At least 1 year without menses and without an alternative medical condition prior to the Screening visit, follicle stimulating hormone FSH levels < 40 mIU/mL and estradiol serum level ≤ 150 pmol/L at Screening
5. Aged at least 18 years but not older than 60 years
6. Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
7. Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)

   Inclusion criteria for SAD, MAD, and FE parts (healthy subjects):
8. Healthy adult male or female
9. Have no clinically significant (CS) diseases captured in the medical history or evidence of CS findings on the physical examination (including vital signs) and/or ECG, as determined by an Investigator

   Inclusion criteria for UC patients:
10. Adult male or female
11. Diagnosis of moderate to severe UC, established at least 6 months prior to Screening; Mayo Score ≥ 6 with rectal bleeding score (RBS) ≥ 1, stool frequency score (SFS) ≥ 1, (mucosal endoscopic score (MES) ≥ 2, and with disease extending ≥ 15 cm from anal verge, and physician's global assessment (PGA)
12. Stable UC symptoms and severity for at least 3 months prior to Screening
13. Well controlled with standard of care therapy for IBD including on stable treatment with aminosalicylates, immunomodulators (eg, methotrexate, azathioprine), or steroids (≤ 20 mg prednisone or equivalent); use of standard of care UC therapies must be stable for at least 4 weeks prior to Screening

Exclusion Criteria:

Exclusion criteria for all subjects and patients:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at Screening or Day -1
3. History of significant hypersensitivity to PALI-2108 or any other PDE4 inhibitor (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability or transit
5. Presence of history of renal disease
6. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease
7. An active infection or a recent history of serious infections in the 30 days prior to first study drug administration
8. Presence of CS vital sign and/or ECG abnormalities (based on the average of triplicate ECG readings) at the Screening visit, as defined by medical judgment
9. Major surgery in the 4 weeks prior to the first study drug administration
10. Vaccination with any live vaccine within 4 weeks prior to study drug administration
11. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
12. Any CS illness in the 28 days prior to the first study drug administration
13. Use of St. John's wort in the 28 days prior to the first study drug administration
14. Any history of tuberculosis
15. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first study drug administration
16. Positive Screening results to HIV antigen/antibody (Ag/Ab) combo, hepatitis B surface antigen, or hepatitis C virus tests
17. Any other CS abnormalities in laboratory test results at Screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
18. Inclusion in a previous group for this clinical study
19. Intake of PALI-2108 in the 28 days prior to the first study drug administration
20. Intake of an investigational drug in the 28 days prior to the first study drug administration
21. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
22. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

    Exclusion criteria for SAD, MAD, and FE parts (healthy subjects):
23. Use of any prescription drugs in the 28 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy
24. Subjects with less than 3 bowel movements or more than 3 episodes of diarrhea (loose watery stools) per week within the month prior to Screening
25. Subjects with history of irritable bowel syndrome and functional dyspepsia

    Exclusion criteria for UC patients:
26. Greater than 2 prior biologic failures
27. Use of a biologic medication within 3 months prior to Screening
28. Use of PDE-4 inhibitors within 3 months prior to Screening
29. History of bariatric surgery, total colectomy with ileorectal anastomosis, or proctocolectomy
30. Presence of a postoperative stoma, ostomy, or ileoanal pouch
31. Participants with any uncontrolled medical conditions, other than active UC, that in the opinion of the Investigator, would put the participant at unacceptable risk or interfere with study assessments or integrity of the data. Other medical conditions should be stable at the time of Screening and be expected to remain stable for the duration of the study
32. Current or history of chronic liver or biliary disease (with the exception of Gilbert's syndrome, asymptomatic gallstones, or uncomplicated fatty liver disease)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAE) or abnormal clinical laboratory measure, electrocardiogram (ECG), or vital sign. [ Safety and Tolerability ] | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 28 ]
  Incidence of Treatment Emergent Adverse Events (TEAE) or abnormal clinical laboratory measure, electrocardiogram (ECG), or vital sign.

SECONDARY OUTCOMES:
Maximum (or peak) plasma concentration (Cmax) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI-2108, PALI-0008, and PALI-0708.
Area Under the Curve from dosing to the time of the last measured concentration (AUC0-T) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI-2108, PALI-0008, and PALI-0708.
Area under the curve from time 0 extrapolated to infinite time (AUCinf) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI-2108, PALI-0008, and PALI-0708.
Time to reach Cmax (Tmax) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI 2108, PALI 0008, and PALI-0708.
Terminal half-life (t1/2) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI 2108, PALI 0008, and PALI-0708.
Ratio of oral clearance (CL/F) (parent only) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI 2108.
Volume of distribution (Vd/F) (parent only) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI 2108.
Ratio of unchanged drug to metabolite (Metabolic ratio) (Cmax) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma Cmax.
Ratio of unchanged drug to metabolite (Metabolic ratio) (AUC) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma AUC.
Concentration of drug and metabolites in feces (C24,f) | MAD and UC Cohort: [ Day 1 to Day 10 ]
  Concentration of PALI-2108, PALI-0708, and PALI-0008 in feces.
Fecal/colonic mucosa drug concentration ratio at steady state (SS). | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  Fecal/colonic mucosa drug concentration ratios of PALI-2108, PALI-0708, and PALI-0008 at Steady State (SS).
Area Under the Curve from dosing to the time of the last measured concentration (AUC0-12) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated in plasma for PALI-2108, PALI-0008, and PALI-0708.
Cumulative drug excreted unchanged in urine (Aetau) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  Cumulative drug excreted unchanged into urine during a dosing interval (Aetau)
Cumulative drug excreted unchanged in urine over 24h (Ae0-24) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  Cumulative drug excreted unchanged in urine over 24h (Ae0-24)
Fraction of drug dose excreted unchanged into urine (fe) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  Fraction of dose excreted unchanged into urine as a percentage (%)
Renal clearance of drug (CLr) (parent only) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  Renal clearance of drug (CLr) of parent only.
Area under the curve from time 0 extrapolated to infinite time (AUC0-12) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI-2108, PALI-0008, and PALI-0708.
Time to last plasma concentration (Tlast) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI-2108, PALI-0008, and PALI-0708.
Terminal rate constant (λz) | SAD and FE Phase: [ Day 1 to Day 7 ], MAD and UC Phase: [ Days 1 to Day 10 ]
  PK parameters calculated for plasma PALI 2108, PALI 0008, and PALI-0708.

OTHER OUTCOMES:
Phosphodiesterase-4 (PDE4)-related pharmacodynamic (PD) biomarkers in MAD and UC | MAD and UC Cohort: [ Day 1 to Day 7 ]
  Mean relative change in Phosphodiesterase-4 (PDE4)-related pharmacodynamic (PD) biomarkers in colon tissue by RNAseq.
Cyclic adenosine monophosphate (cAMP) in MAD and UC | MAD and UC Cohort: [ Day 1 to Day 7 ]
  Mean change from baseline to Day 7 in the concentration of cyclic adenosine monophosphate (cAMP) in colon biopsy tissue.
Colonic tissue drug concentration (Ctissue) in MAD and UC | MAD and UC Cohort: [ Day 1 to Day 7 ]
  Pharmacokinetic (colonic tissue concentration) (Ctissue) of PALI-0008 in colon biopsy.
Mean relative change in microbiome measures in MAD and UC | MAD and UC Cohort: [ Day 1 to Day 10 ]
  Mean change in relative abundance of communities, β-glucuronidase gene, and alpha and beta diversity.
Mean change in fecal calprotectin in UC cohort | UC Cohort: [ Day 1 to Day 10 ]
  Mean change in fecal calprotectin in UC cohort.
Mean change in serum hsCRP in UC cohort | UC Cohort: [ Day 1 to Day 7 ]
  Mean change in serum hsCRP.
Mean change in colon tissue ALC in UC cohort. | UC Cohort: [ Day 1 to Day 7 ]
  Mean change in colon tissue Absolute Lymphocyte Count (ALC) in UC cohort.
Mean change in Nancy Index in UC cohort. | UC Cohort: [ Day 1 to Day 7 ]
  Mean change in Nancy index in UC cohort.
Mean change in Geboes Score in UC cohort. | UC Cohort: [ Day 1 to Day 7 ]
  Mean change in Geboes Score by histopathology n UC cohort.
Mean change in Robart's Histologic Index (RHI) in UC cohort. | UC Cohort: [ Day 1 to Day 7 ]
  Mean change in Robart's Histologic Index (RHI) in UC cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell L Jones, MD, PhD, Principal Investigator — Palisade Bio
Locations (1):
- Altasciences, Montreal, Quebec, Canada